CLINICAL TRIAL: NCT03048500
Title: Parallel Proof of Concept Phase 2 Study of Nivolumab and Metformin Combination Treatment in Advanced Non-small Cell Lung Cancer With and Without Prior Treatment With PD-1/PD-L1 Inhibitors
Brief Title: Nivolumab and Metformin Hydrochloride in Treating Patients With Stage III-IV Non-small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Young Kwang Chae, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16L04; STU00204354 (CTRP (Clinical Trial Reporting Program)); NU 16L04 (Other: Northwestern University); P30CA060553 (NIH); NCI-2017-00060 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage III Non-Small Cell Lung Cancer; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Metformin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (metformin hydrochloride, nivolumab) (Experimental): Patients receive metformin hydrochloride PO once QD on days -7 to -1 and 1-28. Patients also receive nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4, then over 60 minutes on day 1 beginning course 5. Courses repeat every 28 days in the absence of disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Metformin Hydrochloride; Biological: Nivolumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Metformin Hydrochloride — Given PO
  Other Names: Cidophage; Dimefor; Glifage; Glucoformin; Glucophage; Glucophage ER; Metformin HCl; Riomet; Siofor
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
The purpose of this study is to find the benefits of combining nivolumab with metformin in advanced non-small cell lung cancer with and without prior treatment with immunotherapy. We will also be looking at the safety of the combination. Nivolumab is currently approved in certain cancers such as melanoma, lung cancer and kidney cancer. Metformin is approved by the US Food and Drug Administration (FDA) to treat diabetes. In this study, Metformin is being used to treat cancer. This use is not approved by the FDA; therefore, in this study, it is considered experimental. Experimental means the U.S. FDA has not approved the drug for use in your type of cancer. Nivolumab is an antibody (a human protein that sticks to a part of the tumor and/or immune cells) designed to allow the body's immune system to work against tumor cells. It is believed that metformin has immune modifying properties, meaning it can boost your immune system. As a result, it may help certain cancer treatments, known as immunotherapy, to work better.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess anti-tumor activity of the combination treatment of metformin hydrochloride (metformin) with nivolumab in patients with non-small cell lung cancer with and without prior exposure to PD-1/PD-L1 inhibitors.

SECONDARY OBJECTIVES:

I. To assess the efficacy of the combination treatment of metformin with nivolumab according to depth, duration, and persistence of response, disease control rate (DCR; complete response [CR], partial response [PR], and stable disease [SD] at 24 weeks), progression-free survival (PFS), and overall survival (OS) in patients with non-small cell lung cancer with and without prior exposure to PD-1/PD-L1 inhibitors using Response Evaluation Criteria in Solid Tumors (RECIST) criteria version (v)1.1.

II. To assess the efficacy of the combination treatment of metformin with nivolumab according to depth, duration, and persistence of response, objective response rate (ORR), DCR, PFS, and OS in the above population using immune-related RECIST (irRECIST) criteria.

III. To assess the safety and tolerability profile of the combination treatment of metformin with nivolumab in the above population using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

TERTIARY OBJECTIVES:

I. To assess the immune-related tumor and blood biomarkers including T cell markers and their association with treatment response in the above population.

II. To assess the dynamic change in both immune and genomic biomarkers in blood that may correlate with response to metformin.

OUTLINE:

Patients receive metformin hydrochloride orally (PO) once daily (QD) on days -7 to -1 and 1-28. Patients also receive nivolumab intravenously (IV) over 30 minutes on days 1 and 15 of courses 1-4, then over 60 minutes on day 1 beginning course 5. Courses repeat every 28 days in the absence of disease progression, unacceptable toxicity, or withdrawal of consent.

After completion of study treatment, patients are followed up for 30 days, every 3 months for 1 year, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, locally advanced or metastatic stage IV or non-resectable stage III non-small cell lung cancer (NSCLC)
* Patients may have received any number and type of prior treatment regimens for their NSCLC (aside from patients in arm A, who cannot have had PD-1/PD-L1 inhibitors)
* Arm A: patients must be treatment naive to single agent PD-1/PD-L1 inhibitors including but not limited to durvalumab, pembrolizumab, atezolizumab, nivolumab, and avelumab

  * Arm B: patients' tumor must be either refractory to or progressed on one of the above agents
  * Both cases are defined by initial progressive disease (PD) or PD after CR, PR, or SD using RECIST criteria, respectively
* Patients must have measurable disease according to the standard RECIST version 1.1

  * NOTE: computed tomography (CT) scans or magnetic resonance imaging (MRI)s used to assess the measurable disease must have been completed with 28 days prior to the study drug initiation
* Patients need to have adequate kidney, bone marrow, and liver functions =< 14 days of registration as specified below:
* Absolute neutrophil >= 1,000/mcL; transfusion and/or growth factor are permitted within any timeframe
* Platelets >= 50,000/mcl; transfusion and/or growth factor are permitted within any timeframe
* Total bilirubin =< 1.5 times the institutional upper limit of normal (ULN) (or =< 3 times ULN in case of liver metastasis or Gilbert syndrome)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SPGT]) =< 2.5 X institutional ULN (or =< 5 times ULN in case of liver metastasis)
* Creatinine =< 1.4 ng/mL for females; =< 1.5 ng/mL for males; patients with creatinine =< 2.0 ng/mL may still be eligible if in the opinion of the investigator, the benefits of treatment outweigh the risks
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study
* Females of child-bearing potential (FOCBP) and men who are sexually active must agree to follow instructions for method(s) of contraception for the duration of treatment and the designated post-treatment period

  * NOTE: a FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative pregnancy test =< 7 days prior to registration on study
* Patients with known history of central nervous system (CNS) metastases are eligible if CNS disease has been radiographically and neurologically stable for at least 6 weeks prior to study registration and do not require corticosteroids (of any dose) for symptomatic management

  * NOTE: CNS imaging is only required at baseline for patients with known history of CNS metastases
* Patients must have the ability to swallow oral medications
* Patients who are known to be EGFR- or ALK-positive must have received prior EGFR- or ALK-targeted therapy, respectively

  * NOTE: in such cases, documentation of EGFR mutation or ALK translocation status should be provided if available

Exclusion Criteria:

* Both arms: patients should not have received metformin within 6 months prior to registration

  * Arm B: patients who were on metformin while on PD-1/PD-L1 inhibitors are not eligible
* Patients should not have received prior immunotherapies (exception; arm B); they include but are not limited to interleukin-2 and other immune checkpoint antagonist targeting CTLA-4, LAG-3, TIM-3, KIR etc. and/or agonists targeting OX40, ICOS, CD137, etc

  * NOTE: prior cancer vaccine treatments are permitted; for arm B, exposure to single agent PD-1/PD-L1 inhibitors are allowed >= 14 days from registration
* Arm B: patients must not have had prior exposure to combination treatment with PD-1/PD-L1 inhibitors and another systemic treatment

  * NOTE: radiation therapy and surgery do not count as combination treatment
* Patients who are intolerant to PD-1/PD-L1 inhibitors and/or metformin are excluded
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use of duration one month or greater), should be excluded; these include but are not limited to patients with a history of:

  * Immune related neurologic disease
  * Multiple sclerosis
  * Autoimmune (demyelinating) neuropathy
  * Guillain-Barre syndrome
  * Myasthenia gravis
  * Systemic autoimmune disease such as systemic lupus erythematosus (SLE)
  * Connective tissue diseases
  * Scleroderma
  * Inflammatory bowel disease (IBD)
  * Crohn's
  * Ulcerative colitis
  * Patients with a history of toxic epidermal necrolysis (TEN)
  * Stevens-Johnson syndrome
  * Anti-phospholipid syndrome

    * NOTE: subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Patients are ineligible who have any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications =< 14 days prior to registration

  * NOTE: inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; a brief (less than 3 weeks) course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by a contact allergen) is permitted
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Uncontrolled hypertension - blood pressure >= 150/90 mmHg despite medical therapy
  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Patients must not have had another primary malignancy within 2 years prior to starting study treatment with the exception of adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, or in-situ carcinoma of the uterine cervix, or any local cancers that are deemed to be cured from investigator's point of view
* Patients may not be receiving any other investigational agents =< 14 days from registration
* Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) are excluded
* Patients who have any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection are excluded
* Patients with known diabetes whose glucose control or general health condition may be adversely affected by the use of metformin as per the study protocol as deemed by either the study investigator or endocrinologist are excluded
* Patients must not have any of the following contraindications to metformin:

  * Hypersensitivity to metformin or any component of the formulation
  * Kidney dysfunction or abnormal creatinine (Cr < 2 ng/mL) from any cause
  * Acute or metabolic acidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2021-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Young K. Chae, MD, MPH, MBA, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Northwestern University- Lake Forest Hospital, Lake Forest, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient started treatment July 12, 2017. The study was designed to enroll patients with/without prior PD-1/PD-L1 inhibitor treatment. The study closed enrollment to patients without prior treatment with PD-1/PD-L1 inhibitor April 30, 2018. The study was suspended for IA and subsequently closed to further enrollment August 13, 2019.
Groups:
- Treatment (Metformin Hydrochloride, Nivolumab): Induction: Patients receive treatment with metformin monotherapy PO QD on Day -7 to -1.
  Main treatment starting Day 1 of Cycle 1: Patients receive metformin PO QD (Days 1-28 of a 28 days cycle) and nivolumab IV every 14 days (on Days 1 and 15 of a 28 day cycle) for the first 4 cycles and then every 28 days, starting Cycle 5 (Day 1 of a 28 day cycle).
  28 day cycles continue in the absence of disease progression, unacceptable toxicity, or withdrawal of consent.
  Laboratory Biomarker Analysis: Correlative studies
  Metformin Hydrochloride: Given PO
  Nivolumab: Given IV
Period: 2 Cycles of Treatment
Arm/Group | Treatment (Metformin Hydrochloride, Nivolumab)
Started | 17
Attempted 1st Cycle | 17
Attempted 2nd Cycle | 16
Completed | 16
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Reached 1st Response/Continued Treatment
Arm/Group | Treatment (Metformin Hydrochloride, Nivolumab)
Started | 16
Assessed for First Response | 16
Went on to Cycle 3 and Beyond | 9
Completed | 9
Not Completed | 7
Not completed — Progressive Disease | 4
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician decision, Patient PS declining | 1
Period: Follow up for 3 Years
Arm/Group | Treatment (Metformin Hydrochloride, Nivolumab)
Started (All patients that are treated on study go into the follow-up period.) | 16 (1 patient died whilst on study.)
Completed | 0
Not Completed | 16
Not completed — Currently in Follow-up | 4
Not completed — Death | 12

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Metformin Hydrochloride, Nivolumab)
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of Patients With Non-small Cell Lung Cancer Treated With Nivolumab and Metformin Combination Using RECIST 1.1
Description: Anti-tumor activity will be assessed by ORR (defined as the sum of Complete Responses (CR) and/or Partial Responses (PR)) as measured by CT or MRI scan approximately every 8 weeks and assessed by Response Evaluation Criteria in Solid Tumors, RECIST criteria v1.1 using the patients best response to treatment where:
  CR=Disappearance of all lesions PR=At least a 30% decrease in the sum of the diameters of the target lesions, taking as reference the baseline sum diameters
Time Frame: up to a maximum of 24 weeks from start of treatment (Range of cycles that best response was seen was 2-5 cycles of treatment where 1 cycle =28 days)
Population: All patients who received treatment are considered evaluable (even those who did not complete CT scans for RECIST measurement) except those removed from the study for adverse drug reactions.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Metformin Hydrochloride, Nivolumab)
Number analyzed (Participants) | 17
Participants | 1

2. Secondary Outcome: Depth of Response
Description: Depth of response (stable disease or partial response) defined as the change in the sum of the largest tumor diameters per RECIST v1.1 and irRECIST criteria.
Time Frame: 24 weeks from start of treatment
Reporting Status: Not Posted, anticipated posting 2021-02

3. Secondary Outcome: Duration of Response
Description: Duration of response will be evaluated using RECIST v1.1 and irRECIST criteria.
Time Frame: Up to 3 years
Reporting Status: Not Posted

4. Secondary Outcome: Persistence of Response
Description: Persistence of response will be assessed using RECIST v1.1 and irRECIST criteria.
Time Frame: Up to 3 years
Reporting Status: Not Posted

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR will be evaluated using RECIST v1.1 and irRECIST criteria.
Time Frame: 24 weeks from start of treatment
Reporting Status: Not Posted, anticipated posting 2021-02

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS will be assessed using RECIST v1.1 and irRECIST criteria.
Time Frame: At 1 year than at 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival (OS)
Description: OS will be assessed using RECIST v1.1 and irRECIST criteria.
Time Frame: At 1 year than at 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Objective Response Rate (ORR) of Patients With Non-small Cell Lung Cancer Treated With Nivolumab and Metformin Combination Using irRECIST.
Description: Anti-tumor activity will be assessed by ORR (defined as the sum of Complete Responses (CR) and/or Partial Responses (PR)) as measured by CT or MRI scan approximately every 8 weeks and assessed by irRECIST criteria using the patients best response to treatment where:
  CR=Disappearance of all lesions PR=At least a 30% decrease in the sum of the diameters of the target lesions, taking as reference the baseline sum diameters
  But also new measurable lesions are incorporated in the tumor burden, which is used to determine immune-related progressive disease (irPD), immune-related partial response (irPR), and immune-related complete response (irCR). New non-measurable lesions preclude irCR. Under RECST v1.1, there is no confirmation for PD. Under irRECIST, responses and irPDs must be confirmed by consecutive scans at least 4 weeks apart, assuming no clinical deterioration.
Time Frame: up to a maximum of 24 weeks from start of treatment (Range of cycles that best response was seen was 2-6 cycles of treatment where 1 cycle =28 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Metformin Hydrochloride, Nivolumab)
Number analyzed (Participants) | 17
Participants | 2

9. Secondary Outcome: Incidence of Adverse Events
Description: Assess the safety and tolerability of the combination treatment of metformin with nivolumab by evaluating the number, frequency, and severity of adverse events using CTCAE version 4.03.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Day -7 of Induction with Metformin until 30 days post the last dose of treatment (or at time of initiation of new treatment) for a maximum of 14 cycles for any patient (where 1 cycle = 28 days).
Arm/Group | Treatment (Metformin Hydrochloride, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 13/17
Serious Adverse Events (participants affected / at risk) | 8/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Metformin Hydrochloride, Nivolumab) (N=17)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Non-small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — This resulted in death
Constipation (Gastrointestinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) — Patient reported to also have spesis at the same time as the event
Cardiac arrest and subsequent death (Cardiac disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Hemoptysis and acute chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Metformin Hydrochloride, Nivolumab) (N=17)
Anemia (Blood and lymphatic system disorders) | 6
Cardiac arrest (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 9
Flatulence (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 7
Fever (General disorders) | 2
General disorders and administration site conditions - Other, specify (General disorders) | 4
Non-cardiac chest pain (General disorders) | 2
Lung infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
INR increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 2
Lymphocyte count decreased (Investigations) | 7
Lymphocyte count increased (Investigations) | 1
Weight loss (Investigations) | 8
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 2
Hypersomnia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0
Hypertension (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT03048500/Prot_SAP_000.pdf